CLINICAL TRIAL: NCT01021995
Title: Safety and Efficacy of Long-term Treatment With Echinaforce® Over 4 Months
Brief Title: Echinacea Safety Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: A. Vogel AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 920'134
Record Dates: First submitted 2009-11-30; First posted 2009-12-01 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2011-06

CONDITIONS: Infections
Keywords: Safety of Echinacea in comparison to placebo
MeSH Terms: conditions — Infections | interventions — Echinacea extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- echinacea (Experimental)
  Interventions: Drug: echinacea
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: echinacea — drops, 0.9 ml, tid for 4 months
  Arms: echinacea
Drug: placebo — drops, 0.9 ml tid for 4 months
  Arms: placebo

SUMMARY:
Extracts produced from Echinacea purpurea are traditionally used for the prevention and the acute treatment of influenzal infections like the common cold. The aim of this clinical study is to assess clinical safety and efficacy of a treatment with Echinacea in comparison to placebo. 750 healthy subjects with a history of equal or more than 2 cold episodes per year will be recruited during October and November 2009 and will be treated with either Echinacea or placebo over a period of 4 months.

Throughout the study period adverse events (AEs) and adverse drug reactions (AEs with at least a possible causal relation to the treatment) will be recorded.

Common cold related symptoms will be recorded in a daily diary.

ELIGIBILITY:
Inclusion Criteria:

* On average more than 2 cold episodes per year
* Age above 18 years
* Good physical condition
* Signed informed consent

Exclusion Criteria:

* Women without appropriate and effective contraception
* Participation in a clinical trial 30 days prior to this trial
* Pregnant or breast feeding women
* Subjects with pre-existing cold symptoms for more than 24h at inclusion
* Concurrent participation in another clinical trial
* Intake of antimicrobial and/or antiviral medications at inclusion
* Alcohol and/or drug abuse, narcotic drug addiction before and during trial (more than 50 gr and / or 10 cigarettes per day)
* Psychiatric disorders which may influence the results of the trial,
* epilepsy, suicide attempts
* Planned surgical intervention during the trial.
* Serious chronic diseases which influence the absorption, metabolism and the elimination of the investigational product, especially progressive systemic illnesses like tuberculosis, leukaemia,
* collagen disorders and multiple sclerosis
* Known AIDS, HIV-infections and autoimmune diseases
* Known diabetes mellitus (type 1)
* Corticosteroid-treated asthma
* Atopic and allergic subjects (under medicinal treatment)
* Known allergy to plants of the composite family (Asteraceae)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 757 (Actual)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of Adverse Drug Reactions | 4 months

SECONDARY OUTCOMES:
efficacy | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiff School of Biosciences, Cardiff, Wales, United Kingdom